CLINICAL TRIAL: NCT02951689
Title: Influence of Probiotics on Body Composition and Health in Occupational Shift Workers
Brief Title: Probiotics in Occupational Shift Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Strength and Conditioning Association (Other); Winclove Probiotics B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 16-1397
Record Dates: First submitted 2016-10-27; First posted 2016-11-01 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Shift-Work Related Sleep Disturbance; Healthy
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental): Multi-strain probiotic
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Maltodextrin placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic
  Arms: Probiotic
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Purpose: To evaluate the influence of probiotic supplementation on body composition and other markers of health in occupational shift-workers.

Participants: Healthy, overweight females (ages 22-55 yrs) who are employed on a shift-working schedule.

Procedures (methods): In a randomized, placebo-controlled intervention, subjects will complete 3 different testing sessions (pre-screening, 1 baseline, 1 post-testing session) as well as a 6-week intervention period. Prescreening will include written informed consent, a health history questionnaire, baseline anthropometric measures, assessment of resting heart rate, and exercise protocol familiarization. Baseline testing will involve body composition, a fasted blood draw, mood surveys, and an exercise treadmill test. Subjects will be randomized to a treatment group (multi-strain probiotic or placebo) for 6 weeks of supplementation that includes 2 electronic contacts, followed by post-testing that will occur in the same fashion as baseline testing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, pre-menopausal women
* Currently employed on a shift-working (rotating, evening, or night) schedule and has maintained this schedule ≥ 6 months prior to enrollment
* Participant agrees to maintain usual activity lifestyle
* Participant has a body mass index of ≥25 kg/m2
* Participant has provided written and dated informed consent to participate in the study
* Participant is willing and able to comply with the protocol
* Participant is apparently healthy and free from disease, as determined by a health history questionnaire
* Participant agrees to abstain from smoking, caffeine, tobacco, and alcohol before testing days
* Participant is not currently pregnant and does not desire to become pregnant in the next 8 weeks.

Exclusion Criteria:

* Having a history of medical or surgical events that may significantly affect the study outcome, including cardiovascular disease, metabolic, renal, hepatic, or musculoskeletal disorders
* Participant is using, or has used a probiotic supplements within 8 weeks prior to enrollment
* Participant has lost or gained greater than 8 pounds within the previous 2 months
* Participant is in, or has participated in another clinical trial within 4 weeks prior to enrollment
* Participant had or currently has a self-identified eating disorder
* Participant is pregnant or plans on becoming pregnant
* Participant has a known allergy or sensitivity to any ingredient in the test product or placebo (determined from health history questionnaire)

Ages: 22 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-09; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Visceral Fat | 6 weeks
  measured by ultrasound

SECONDARY OUTCOMES:
Ratio of fat in the abdominal region vs. hip region | 6 weeks
  Measured from dual energy x-ray absorptiometry
Body Fat | 6 weeks
  measured from dual energy x-ray absorptiometry
Lean body mass | 6 weeks
  measured from dual energy x-ray absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: Abbie Smith-Ryan, PhD, Study Director — University of North Carolina, Chapel Hill
Locations (1):
- Applied Physiology Laboratory, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No